CLINICAL TRIAL: NCT02061774
Title: Postoperative Opioid Use and Pain Scores in Patients Undergoing Transforaminal Lumbar Interbody Fusion After Administration of Preoperative Followed by Scheduled Intravenous Acetaminophen:
Brief Title: Postoperative Opioid Use and Pain Scores in Patients Undergoing Transforaminal Lumbar Interbody Fusion
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Preliminary analysis showed not clinically significant. Study ended and closed 1/11/2018
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L14-015
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Low Back Pain
Keywords: acetaminophen in transforaminal lumbar interbody fusion
MeSH Terms: conditions — Low Back Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- acetaminophen (Active Comparator): 1g intravenous acetaminophen over a period of 15 minutes, 15 minutes (+/- 10 minutes) prior to the anticipated time of incision and every 6 hours (+/- 30 minutes) after the initial dose for 24 hours; maximum dose of 4 grams in 24 hours
  Interventions: Drug: Acetaminophen
- PlaceboComparator (Placebo Comparator): Placebo Comparator 0.9% NaCl 100 mL over will be administered intravenously over a period of 15 minutes, 15 minutes (+/- 10 minutes) prior to the anticipated time of incision and every 6 hours (+/- 30 minutes) after the initial dose for 24 hours
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Acetaminophen — 1 gram of intravenous Acetaminophen
  Other Names: Tylenol
  Arms: acetaminophen
Drug: Placebo comparator — placebo comparator .9% NaCl (sodium chloride) 100 mL over will be administered intravenously over a period of 15 minutes, 15 minutes (+/- 10 minutes) prior to the anticipated time of incision and every 6 hours (+/- 30 minutes) after the initial dose for 24 hours
  Other Names: placebo
  Arms: PlaceboComparator

SUMMARY:
The purpose of this project is to study the effects of preoperative followed by scheduled intravenous acetaminophen on pain control for 24 hours postoperatively after minimally invasive 1 or 2 level transforaminal lumbar interbody fusion.

DETAILED DESCRIPTION:
The purpose of this project is to study the effects of preoperative followed by scheduled intravenous acetaminophen on pain control for 24 hours postoperatively after minimally invasive 1 or 2 level transforaminal lumbar interbody fusion. The advantages of intravenous acetaminophen are well known in the literature and its opioid-sparing effects have been documented in multiple surgical studies.

Multimodal regimens are now being advocated in the literature to decrease opioid use (8, 23). This is especially significant in spine surgery patients who often have chronic pain requiring long-term use of these habit-forming drugs as well as in patients who may not be able to tolerate opiods due to health status.

To our knowledge there are no studies done in the U.S. on the opioid sparing and pain reducing effects of intravenous acetaminophen on patients undergoing elective minimally invasive 1 or 2 level transforaminal lumbar interbody fusion. Investigating intravenous acetaminophen, particularly its pain reducing and opioid sparing effects, may give surgeons another medication for use in a multimodal approach to pain.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Being scheduled to have elective primary minimally invasive 1 or 2 level transforaminal lumbar laminectomy interbody fusion
* ASA I, II, or III
* Informed consent form signed

Exclusion Criteria:

* Anyone weighing less than 50kg (as this would require a dosing change).
* Hypersensitivity or contraindication to intravenous acetaminophen or opioids
* Allergy to Methocarbamol; morphine sulfate, sevoflourane, or fentanyl
* Impairment of liver function-- defined as the inability to receive intravenous acetaminophen without dose adjustment as determined by the investigator; or history of chronic liver disease defined as history of hepatitis of any kind as recorded in the patient's chart
* Mental retardation recorded as a diagnosis in the patient's chart
* History of chronic pain (defined as currently receiving treatment from a specialist for pain)
* History of pain recalcitrant to intravenous morphine
* Impaired kidney function (defined as creatinine > 1.5)
* Anyone who is not a candidate for general anesthesia or any other portion of the investigator's standard of

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10; Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Felton, MD, Principal Investigator — TTUHSC department of Surgery
Locations (1):
- Texas Tech University Health Science Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acetaminophen | PlaceboComparator
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | PlaceboComparator | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 54.5 [44 to 61] | 54.0 [51 to 61] | 54.5 [44 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21
ASA score [Number; unit: participants] — ASA I A normal healthy patient, ASA II A patient with mild systemic disease. Mild diseases only without substantive functional limitations.
  ASA III A patient with severe systemic disease Substantive functional limitations; One or more moderate to severe diseases.
  ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
  participants
    ASA 1 | 1 | 1 | 2
    ASA 2 | 6 | 5 | 11
    ASA 3 | 3 | 4 | 7
decompressions [Count of Participants; unit: Participants]
  1 decompression | 9 | 9 | 18
  2 decompressions | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: VAS
Description: The Visual Analogue Scale (VAS) and Verbal Rating Scale (VRS) will be measured at 4 hour intervals for a 24-hr period - measures of pain intensity in clinical and research settings. 0-10 Numeric pain intensity scale. 0 is no pain, 5 is moderate pain, and 10 is worst possible pain
Time Frame: Q4 x 24 hours averaged
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Acetaminophen | PlaceboComparator
Number analyzed (Participants) | 10 | 11
score on a scale | 6 [4 to 7.2] | 8.5 [4.8 to 10.0]

2. Secondary Outcome: Level of 100% Sedation
Description: Sedation will be measured on a scale of 1 to 5 at 4-hour intervals as follows: 1-completely awake; 2-awake but drowsy; 3 asleep, but responds to verbal commands; 4-asleep but responds to tactile stimuli; and 5-asleep and not responding to any stimuli.
Time Frame: 4-hr intervals for a 24-hr period averaged
Measure: Number; unit: participants of 100% sedation
Arm/Group | Acetaminophen | PlaceboComparator
Number analyzed (Participants) | 10 | 11
participants of 100% sedation | 10 | 11

3. Secondary Outcome: Vital Signs
Description: Routine postoperative vital signs will be collected at 4-hour intervals (+/- 30 minutes) postoperatively respiratory rate, oxygen saturation, mean arterial pressure, and heart rate. Any reports of headache, dizziness, nausea, vomiting, pruritis, agitation, constipation, insomnia, bradycardia (Heart rate below 60 beats per minute), hypotension (MAP less than 30% of baseline), or urinary retention will be recorded throughout the study and will be treated appropriately as they occur, and the treatment medication will be stopped if determined to be a causative factor.
Time Frame: 4-hour intervals (+/- 30 minutes) for 24-hrs averaged
Measure: Number; unit: participants with 100% vitals completed
Arm/Group | Acetaminophen | PlaceboComparator
Number analyzed (Participants) | 10 | 11
participants with 100% vitals completed | 10 | 11

4. Other Pre Specified Outcome: Total PCA Morphine
Description: Amount of morphine used during surgery
Time Frame: Duration of operation
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Acetaminophen | PlaceboComparator
Number analyzed (Participants) | 10 | 11
mg | 41.6 [29 to 67.5] | 36.6 [26 to 55.3]

ADVERSE EVENTS:
Time Frame: 6 months
Description: adverse event information does not differs from the clinicaltrials.gov defination
Arm/Group | Acetaminophen | PlaceboComparator
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

LIMITATIONS AND CAVEATS:
Early Termination due to preliminary analysis showed not clinically significant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT02061774/Prot_SAP_000.pdf